CLINICAL TRIAL: NCT00467714
Title: Evaluation of Cloumella Strut in Maintenance of Tip Rotation
Brief Title: Evaluation Of Cloumella Strut Effect In Tip Rotation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: tums.ac.ir, ENT research center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BS-181351
Record Dates: First submitted 2007-04-29; First posted 2007-05-01 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-11

CONDITIONS: Nose Deformities, Acquired
Keywords: RHINOPLASTY ,ESTHETIC SURGERY
MeSH Terms: conditions — Nose Deformities, Acquired | interventions — Rhinoplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (No Intervention): 2.5 cm Cartilage as columella strut
  Interventions: Procedure: rhinoplasty

INTERVENTIONS:
Procedure: rhinoplasty — COLUMELLA STRUT PLACEMENT
  Other Names: no other name

SUMMARY:
The role of strut in rhinoplasty has been debated for many years and many research has been made over this problem but there is no significant data for descision of surgeon, so this study was designed to evaluate the effect of columellar strut in tip projection and rotation.

DETAILED DESCRIPTION:
In selected case of rhinoplasty use strut randomly and blindly evalute the effect of it in tip rotation and projection.

ELIGIBILITY:
Inclusion Criteria:

* RHINOPLASTIC PATIENTS

Exclusion Criteria:

* REVISION SURGERY,
* INCOMPLETE STRIP,
* FACIAL ANOMALY

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
TIP ROTATION | 6 month after surgery

SECONDARY OUTCOMES:
TIP PROJECTION | 6 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: mohmad sadeghi, professor, Study Director — deputy of research of tehran university medical science
Locations (1):
- Imam Hospital, Tehran, Tehran Province, Iran